CLINICAL TRIAL: NCT00390819
Title: Epidemiology of Community Acquired Pneumonia in North Israel
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: HaEmek Medical Center, Israel (Other)
Other Study IDs: 131074
Record Dates: First submitted 2006-10-19; First posted 2006-10-20 (Estimated); Last update posted 2006-10-20 (Estimated); Status verified 2006-10

CONDITIONS: Community Acquired Pneumonia
Keywords: Community acquired pneumonia
MeSH Terms: conditions — Community-Acquired Pneumonia

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

SUMMARY:
Pneumonia in general and CAP in particular is considered as one of the most common bacterial infections, associated with high rates of morbidity and mortality and is highly significant economically since all respiratory infections, and pneumonia especially, cause about 80% of antimicrobials use in the community. The high frequency of respiratory infections and the excessive use of antimicrobials are major contributors to the development of pathogens resistant to antimicrobials. In addition, in CAP almost all patients are treated empirically, without identification of causing pathogen.

Aim of study: To identify common pathogens causing CAP in hospitalized patients in north Israel.

DETAILED DESCRIPTION:
Pneumonia in general and CAP in particular is considered as one of the most common bacterial infections, associated with high rates of morbidity and mortality.

CAP is highly significant economically since all respiratory infections, and pneumonia especially, cause about 80% of antimicrobials use in the community. The high frequency of respiratory infections and the excessive use of antimicrobials are major contributors to the development of pathogens resistant to antimicrobials. In addition, in CAP almost all patients are treated empirically, without identification of causing pathogen.

CAP is divided to two principal groups: Bacterial CAP and Atypical CAP. Since pathogens are different, treatment approach is also different. The main obstacle is absence of adequate diagnostic immediate and cheap tools to enable identifying pathogen and hence treatment is not always appropriate. Giving the right therapy at the right time is of major importance since early start of correct treatment is linked to morbidity and mortality of patients. For prescribing appropriate empiric therapy, knowing the epidemiology of CAP, i.e. the frequent causing pathogens according to age groups and other demographic characteristics, is essential.

Unfortunately, except one study conducted 10 years ago by Dr. Liberman from Soroka Medical Center, there is no characteristic information regarding causing pathogens. Lacking this data, might result in selecting inadequate treatment.

Material & Methods:

We should enroll about 300 patients hospitalized in Ha'Emek Medical Center with the diagnosis of CAP, in order to make the study results statistically significant.

In addition to demographic and clinical data, following tests will be performed:

1. Blood cultures
2. Sputum
3. PCR - throat culture to the following pathogens:

   * Mycoplasma pneumoniae
   * Chlamydia pneumoniae
   * Legionella
   * Adenovirus
   * Influenza A
   * Influenza B
   * RSV
   * Metapneumovirus
   * Parainfluenza
   * Pneumococcal antigen in urine

ELIGIBILITY:
Inclusion Criteria:

* Community acquired pneumonia
* Hospitalization

Exclusion Criteria:

* Immunocompromised patients
* Patients under chemotherapy treatment
* Patients under steroids treament

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2006-11

CONTACTS AND LOCATIONS:
Overall Officials: Fahmi Shibli, M.D., Principal Investigator — Ha'Emek Medical Center, Afula, Israel
Locations (1):
- Ha'Emek Medical Center, Afula, Israel

REFERENCES:
- [Background] Porath A, Schlaeffer F, Lieberman D. The epidemiology of community-acquired pneumonia among hospitalized adults. J Infect. 1997 Jan;34(1):41-8. doi: 10.1016/s0163-4453(97)80008-4. PMID 9120323